CLINICAL TRIAL: NCT01600066
Title: Erectile Dysfunction in Severe Obstructive Sleep Apnea : Effects of CPAP Therapy
Brief Title: Erectile Dysfunction in Severe Obstructive Sleep Apnea: Effects of CPAP Therapy
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Richard Schulz, Prof. Dr. Richard Schulz, University of Giessen
Other Study IDs: GERSAN-1; UGLC (Other: UGLC)
Record Dates: First submitted 2012-05-09; First posted 2012-05-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Obstructive Sleep Apnea; Erectile Dysfunction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimens for the determination of lipids and glucose
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Obstructive sleep apnea has been linked to erectile dysfunction. Furthermore, small studies suggest that treatment of sleep apnea by continuous positive airway pressure (CPAP) may reverse erectile dysfunction in affected patients. The present study aims to investigate in a larger cohort if severe sleep apnea is independently associated with erectile dysfunction and if 6-12 months of CPAP therapy lead to an improvement of erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* apnea-hypopnea-index > 30/h
* no CPAP therapy
* male gender
* 18-80 years of age
* having or attempting to have regular sexual intercourse

Exclusion Criteria:

* apnea-hypopnea-index < 30/h
* already treated by CPAP
* female gender
* age < 18 or > 80 years
* not having or not attempting to have regular sexual intercourse

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male patients with untreated severe sleep apnea (apnea-hypopnea-index > 30/h)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of erectile function in severe sleep apnea after 6-12 months of CPAP therapy | at the time of diagnosis of sleep apnea and after 6-12 months of CPAP therapy
  an established self-administered questionnaire is used to assess changes in erectile function occurring after 6-12 months of CPAP therapy in patients with severe sleep apnea

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schulz, MD, Principal Investigator — University of Giessen Lung Center, Germany